CLINICAL TRIAL: NCT06715358
Title: Cluster Randomized Trial for the SI! Program Reintervention for Elementary Schools
Brief Title: The SI! Program Reintervention for Elementary Schools Trial
Acronym: PSIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Science, Health and Education, Spain (Other)
Collaborators: La Caixa Foundation (Other); Centro Nacional de Investigaciones Cardiovasculares Carlos III (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHE-004-SI
Record Dates: First submitted 2024-11-19; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Health; Obesity
Keywords: Cardiovascular health; Health promotion; School-based intervention; Children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reintervention (Active Comparator): Implement the SI! Program environment intervention from 2nd grade throughout the whole Elementary Education (5 years) and with two classroom interventions: one at 2nd grade and a reintervention at 5th grade.
  Interventions: Behavioral: Reintervention
- Late intervention (Active Comparator): Implement the SI! Program environment intervention from 5th grade throughout the rest of the Elementary Education (2 years) with only one classroom intervention at 5th grade.
  Interventions: Behavioral: Late intervention

INTERVENTIONS:
Behavioral: Reintervention — * SI! Program environment intervention from 2nd grade through all Elementary Education.
  * SI! Program classroom intervention in 2nd grade.
  * SI! Program classroom intervention in 5th grade.
  Arms: Reintervention
Behavioral: Late intervention — * SI! Program environment intervention from 5th grade through all Elementary Education.
  * SI! Program classroom intervention in 5th grade.
  Arms: Late intervention

SUMMARY:
Background and objectives:

The SI! Program is a multilevel school-based intervention that has been previously evaluated in different ages in three countries. Schools were randomized to the SI! Program intervention or the control group, and prior to and after the intervention several questionnaires and direct measures were used to assess changes in lifestyle and cardiovascular health indicators. In the SI! Program for Preschool, children in the intervention group increased significantly more their knowledge, attitudes and habits after 4 months of the implementation of the SI! Program compared to children in the control group. However, until now, results have shown that improvements in cardiovascular health between 3 and 5 years old do not sustain overtime. For this reason, the new project of the SI! Program proposes a reinforcement of the children's environment to boost the effect of the intervention and a reinforcement in the classroom after 2 years to favor the sustainability of the effect. The main objective of this study is to assess the effect of the reintervention of the SI! Program in the SI!-Child health score in Elementary school children (7-12 years old) and compare its effect with a single late exposure to the SI! Program.

Methodology:

A cluster-randomized trial involving 50 elementary schools in Spain will be carried out. Schools will be 1:1 randomized to either implement the SI! Program from 2nd grade throughout the whole Elementary Education (5 years) with two classroom interventions (one at 2nd grade and one at 5th grade) or to implement the SI! Program from 5th grade throughout the rest of the Elementary Education (2 years) with only one classroom intervention at 5th grade. Children in the first year of Elementary education at the beginning of the trial will be recruited. Participants will be evaluated at baseline, and after 3, 5 and 6 years using a battery of measurements on cardiovascular health parameters (anthropometry, bioimpedance, blood analysis, accelerometers, questionnaires). The primary endpoint will be the change in the SI!-Child score after 5 years. The SI! Child score includes sleep, diet, physical activity and nutritional status, and ranges from 0 to 100, with higher scores indicating better cardiovascular profiles. Secondary outcomes include the change in individual components of the SI!-Child score and other cardiovascular health indicators such as sedentarism, tobacco exposure, adiposity, blood pressure, lipid profile and blood glucose, and to assess the effect of the SI! Program reintervention to maintain or improve all cardiovascular health indicators previously mentioned one year after the reintervention.

Expected results:

The investigators expect to show that a school-based educational intervention with a reinforcement in the classroom after 2 years in addition to a school environment intervention will induce favorable and sustainable lifestyle changes in health behaviors among Spanish children. If successful, this strategy could be widely adopted having a meaningful effect on cardiovascular health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Schools from the Madrid Region or Catalonia.
* Public or charter schools
* Schools having from 1st to 6th grades and at least one classroom in 1st grade.
* Schools having a canteen
* Children in the 1st grade.

Exclusion Criteria:

* None

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Change in the SI!-Child health score at the end of the intervention | From baseline assessment to the end of the intervention, an average of 5 years
  The primary outcome will be the difference in the SI!-Child score (0-100 points for each component, higher scores indicating healthier habits) between the reintervention group and the late intervention group. The SI! Child score includes Sleep (measured as hours of sleep), Diet (fruits and vegetables, sugared beverages, fast-food, legumes and nuts, sweets and pastries), Physical activity (minutes of moderate and vigorous physical activity), Nutritional status (body mass index calculated as body weight divided by height squared (kg/m2).

SECONDARY OUTCOMES:
Effect of the SI! Program reintervention in the individual components of the SI!-Child health score | From baseline assessment to the end of the intervention, an average of 5 years
  Mean score and change at follow-up visits for each of the individual components of the SI! Child score (0-100 points for each component, higher scores indicating healthier habits): Sleep (measured as hours of sleep ), Diet (fruits and vegetables, sugared beverages, fast-food, legumes and nuts, sweets and pastries), Physical activity (minutes of moderate and vigorous physical activity), nutritional status (body mass index calculated as body weight divided by height squared (kg/m2)).

OTHER OUTCOMES:
Effect of the SI! Program reintervention in sedentary time | From baseline assessment to the end of the intervention, an average of 5 years
  Mean and change in minutes of sedentary time assessed with a wrist-worn Actigraph wGT3X-BT accelerometer.
Effect of the SI! Program reintervention in screen time | From baseline assessment to the end of the intervention, an average of 5 years
  Mean and change in hours of screen time assessed with a specific questionnaire asking the number of hours of leisure and non-leisure screen time during the week and during the weekends.
Effect of the SI! Program reintervention in tobacco exposure | From baseline assessment to the end of the intervention, an average of 5 years
  Prevalence and change in tobacco exposure assessed with a direct question asking if anyone who lives with the child smokes (binary variable of yes/no).
Effect of the SI! Program reintervention in body mass index | From baseline assessment to the end of the intervention, an average of 5 years
  Mean and change in body mass index (calculated as body weight divided by height squared (kg/m2)). Body height as measured using a stadiometer (Seca 213). Body weight as measured using the OMRON BF511 electronic scale.
Effect of the SI! Program reintervention in waist circumference | From baseline assessment to the end of the intervention, an average of 5 years
  Mean and change in waist circumference (cm). Waist circumference as measured using a Holtain tape.
Effect of the SI! Program reintervention in blood pressure | From baseline assessment to the end of the intervention, an average of 5 years
  Mean and change in blood pressure (systolic and diastolic) (mmHg) as assessed with a fully automated blood pressure monitor (OMRON M6 monitor).
Effect of the SI! Program reintervention in the lipid profile and blood glucose levels | From baseline assessment to the end of the intervention, an average of 5 years
  Mean total, LDL- and HDL-cholesterol (mg/dL), and blood glucose (mg/dL) and change at follow-up visits as evaluated by point-of-care testing. Blood glucose and lipid profile were measured using a CardioCheck Plus device and PTS-Panels test strips in capillary blood sampled with a lancet in fasting status.
Change in the SI!-Child score one year after the intervention | From baseline assessment to the end of the trial, an average of 6 years
  Differences one year after the reintervention (~13 years of age) in the SI!-Child score (0-100 points for each component, higher scores indicating healthier habits): Sleep (measured as hours of sleep), Diet (fruits and vegetables, sugared beverages, fast-food, legumes and nuts, sweets and pastries), Physical activity (minutes of moderate and vigorous physical activity), Nutritional status (body mass index calculated as body weight divided by height squared (kg/m2).

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, Principal Investigator — Mount Sinaí Hospital
Locations (1):
- Foundation for Science, Health and Education, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request, with the approval of the Steering Committee and the signing of a data exchange agreement.
Time Frame: 9 months after publication
Access Criteria: The de-identified data underlying results in a publication will be shared on reasonable request to the principal investigator.
  Email: estudio@fundacionshe.org
URL: https://fundacionshe.org/programa-si

REFERENCES:
- [Background] Penalvo JL, Sotos-Prieto M, Santos-Beneit G, Pocock S, Redondo J, Fuster V. The Program SI! intervention for enhancing a healthy lifestyle in preschoolers: first results from a cluster randomized trial. BMC Public Health. 2013 Dec 20;13:1208. doi: 10.1186/1471-2458-13-1208. PMID 24359285
- [Background] Penalvo JL, Santos-Beneit G, Sotos-Prieto M, Martinez R, Rodriguez C, Franco M, Lopez-Romero P, Pocock S, Redondo J, Fuster V. A cluster randomized trial to evaluate the efficacy of a school-based behavioral intervention for health promotion among children aged 3 to 5. BMC Public Health. 2013 Jul 15;13:656. doi: 10.1186/1471-2458-13-656. PMID 23855415
- [Background] Penalvo JL, Santos-Beneit G, Sotos-Prieto M, Bodega P, Oliva B, Orrit X, Rodriguez C, Fernandez-Alvira JM, Redondo J, Vedanthan R, Bansilal S, Gomez E, Fuster V. The SI! Program for Cardiovascular Health Promotion in Early Childhood: A Cluster-Randomized Trial. J Am Coll Cardiol. 2015 Oct 6;66(14):1525-1534. doi: 10.1016/j.jacc.2015.08.014. PMID 26429075
- [Background] Santos-Beneit G, Bodega P, de Miguel M, Rodriguez C, Carral V, Orrit X, Haro D, Carvajal I, de Cos-Gandoy A, Penalvo JL, Gomez-Pardo E, Oliva B, Ibanez B, Fernandez-Alvira JM, Fernandez-Jimenez R, Fuster V. Rationale and design of the SI! Program for health promotion in elementary students aged 6 to 11 years: A cluster randomized trial. Am Heart J. 2019 Apr;210:9-17. doi: 10.1016/j.ahj.2018.12.011. Epub 2019 Jan 8. PMID 30716509
- [Background] Fernandez-Jimenez R, Santos-Beneit G, Tresserra-Rimbau A, Bodega P, de Miguel M, de Cos-Gandoy A, Rodriguez C, Carral V, Orrit X, Haro D, Carvajal I, Ibanez B, Storniolo C, Domenech M, Estruch R, Fernandez-Alvira JM, Lamuela-Raventos RM, Fuster V. Rationale and design of the school-based SI! Program to face obesity and promote health among Spanish adolescents: A cluster-randomized controlled trial. Am Heart J. 2019 Sep;215:27-40. doi: 10.1016/j.ahj.2019.03.014. Epub 2019 Apr 10. PMID 31277052
- [Background] Santos-Beneit G, Fernandez-Jimenez R, de Cos-Gandoy A, Rodriguez C, Carral V, Bodega P, de Miguel M, Orrit X, Haro D, Penalvo JL, Fernandez-Alvira JM, Peyra C, Cespedes JA, Turco A, Hunn M, Jaslow R, Baxter J, Carvajal I, Fuster V. Lessons Learned From 10 Years of Preschool Intervention for Health Promotion: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Jan 25;79(3):283-298. doi: 10.1016/j.jacc.2021.10.046. PMID 35057915
- [Background] Santos-Beneit G, Fernandez-Alvira JM, Tresserra-Rimbau A, Bodega P, de Cos-Gandoy A, de Miguel M, Ramirez-Garza SL, Laveriano-Santos EP, Arancibia-Riveros C, Carral V, Orrit X, Rodriguez C, Carvajal I, Haro D, Peyra C, Martinez-Gomez J, Alvarez-Benavides A, Estruch R, Lamuela-Raventos RM, Fernandez-Jimenez R, Fuster V. School-Based Cardiovascular Health Promotion in Adolescents: A Cluster Randomized Clinical Trial. JAMA Cardiol. 2023 Sep 1;8(9):816-824. doi: 10.1001/jamacardio.2023.2231. PMID 37531100
- [Background] Santos-Beneit G, Bodega P, de Cos-Gandoy A, de Miguel M, Rodriguez C, Orrit X, Carral V, Haro D, Carvajal I, Peyra C, Martinez-Gomez J, Fernandez-Alvira JM, Fernandez-Jimenez R, Fuster V. Effect of Time-Varying Exposure to School-Based Health Promotion on Adiposity in Childhood. J Am Coll Cardiol. 2024 Aug 6;84(6):499-508. doi: 10.1016/j.jacc.2024.04.065. PMID 39084824
- See also: Web of the SHE Foundation — https://fundacionshe.org/
- See also: Web of the SI! Program — https://fundacionshe.org/en/si-program/